CLINICAL TRIAL: NCT02958085
Title: Investigation of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Dosing of NNC0174-0833 in Subjects With Obesity or Overweight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN9838-4021; U1111-1131-7209 (Other: WHO)
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NNC0174-0833 (Experimental)
  Interventions: Drug: NNC0174-0833
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0174-0833 — Doses of NNC0174-0833, dosed either once daily or once weekly
  Arms: NNC0174-0833
Drug: Placebo — Dosed either once daily or once weekly
  Arms: Placebo

SUMMARY:
This trial is conducted in The United States of America. The aim of this trial is to investigate Safety, Tolerability, Pharmacokinetics (the exposure of the trial drug in the body) and Pharmacodynamics (the effect of the investigated drug on the body) of Multiple Dosing of NNC0174-0833 in Subjects with Obesity or Overweight.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential (NCBP), aged 22-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 25.0 and 39.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess of adipose tissue, as judged by the investigator

Exclusion Criteria:

* History or presence of any clinically relevant respiratory, metabolic, renal, hepatic,gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or other major disorders including sleep apnoea or excessive sleepiness that might require medical attention
* History or presence of cardiovascular disease including stable and unstable angina, myocardial infarction, transient ischaemic attack, stroke, cardiac decompensation, and heart failure
* History or presence of a disease being associated with impaired calcium homeostasis and/or increased bone turnover (e.g. Paget´s disease, osteoporosis)
* Male subject who is not surgically sterilised (vasectomy) and is sexually active with female partner(s) and is not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their non-pregnant female partner(s) of childbearing potential (Pearl Index below 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide), and/or intend to donate sperm in the period from screening until 3 months following administration of the last dose of investigational medical product

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From time of first dosing (Day 1) to the post-treatment follow-up visit (Day 99)

SECONDARY OUTCOMES:
The area under the NNC0174-0833 plasma concentration-time curve | From time 0 to 24 hours at steady state
  [only applicable for once daily dosing]
The area under the NNC0174-0833 plasma concentration-time curve | From time 0 to 168 hours at steady state
  [only applicable for once weekly dosing]
The maximum concentration of NNC0174-0833 in plasma at steady state | Day 1; Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Overland Park, Kansas, United States